CLINICAL TRIAL: NCT01812395
Title: Is Superior Laryngeal Nerve Really Safe During Thyroidectomy Using Ultrasonic Dissector.
Brief Title: Thyroidectomy Using Ultrasonic Dissector: Is Superior Laryngeal Nerve Really Safe ?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: S.B. Konya Education and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KEAH07031301; U1111-1140-3809 (Other: WHO Universal Trial Number)
Record Dates: First submitted 2013-03-08; First posted 2013-03-18 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Goiter
Keywords: thyroidectomy; ultrasonic dissector; harmonic focus device; superior laryngeal nerve
MeSH Terms: conditions — Goiter

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasonic Dissector Thyroidectomy (Active Comparator): Thyroidectomy using harmonic focus (r) device
  Interventions: Device: Thyroidectomy using harmonic focus (r)
- Classic thyroidectomy (Active Comparator): Patients having conventional thyroidectomy
  Interventions: Procedure: Conventional thyroidectomy

INTERVENTIONS:
Device: Thyroidectomy using harmonic focus (r) — Harmonic focus(r) device is used to seal and cut the vessels during thyroidectomy.
  Other Names: Ethicon(r) Harmonic Focus(r) Curved Shears
  Arms: Ultrasonic Dissector Thyroidectomy
Procedure: Conventional thyroidectomy — Vessels are ligated with sutures then cut using classic scalpel or scissors.
  Arms: Classic thyroidectomy

SUMMARY:
New devices and techniques are coming into use everyday. Ultrasonic dissectors (UDs) are such new devices which is a practical alternative to the usage of scalpel and sutures. UD's cause overheating of neighboring tissues in an area of 1 to 3 millimeters. Due to the generated heat UDs might cause nerve injury. The investigators would like to see if usage of UDs during thyroidectomy poses a risk for superior laryngeal nerve injury compared to conventional thyroidectomy.

DETAILED DESCRIPTION:
We see new advances in the practice of surgery nearly everyday. New techniques and devices became available and even newer ones are under developement. Ultrasonic Dissectors (UDs) which are primarily developed for laparoscopic surgery found widespread use in thyroid surgery. UDs while closing the nearby vessels cause overheating of neighboring tissues in a 1-3 mm. area. Due to the generated heat UDs might cause nerve injury. We would like to see if usage of UDs during thyroidectomy poses a risk for superior laryngeal nerve injury compared to conventional thyroidectomy where vessels are first sealed with sutures then cut. To this end patients in both conventional and ultrasonic dissector thyroidectomy arms will be checked for superior laryngeal nerve function the day following operation and six months later.

ELIGIBILITY:
Inclusion Criteria:

* Patients having thyroidectomy

Exclusion Criteria:

* Previous neck surgery
* Thyroid cancers
* History of superior or inferior laryngeal nerve paralysis
* History of neck irradiation
* Pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of superior laryngeal nerve function | 6 months
  Patients will be checked for superior laryngeal nerve function by laryngostroboscopy one day after thyroidectomy and 6 months after thyroidectomy.

SECONDARY OUTCOMES:
Assessment of inferior laryngeal nerve function | 6 months
  Patients will be checked for inferior laryngeal nerve function by laryngostroboscopy one day after thyroidectomy and 6 months after thyroidectomy.
Assessment of other complications | 1 week
  Whether patients develop postoperative seroma, haematoma, infection or maceration will be recorded

OTHER OUTCOMES:
Assessment of hemorrhage | 3 day
  Amounts of peroperative and postoperative hemorrhage will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Osman DOĞRU, M.D., Study Director — Konya Education and Research Hospital General Surgery Clinic
Locations (1):
- Konya Education and Research Hospital, Meram, Konya, Turkey (Türkiye)

REFERENCES:
- [Background] Pardal-Refoyo JL. [Hemostatic systems in thyroid surgery and complications]. Acta Otorrinolaringol Esp. 2011 Sep-Oct;62(5):339-46. doi: 10.1016/j.otorri.2011.03.004. Epub 2011 May 6. Spanish. PMID 21529721
- [Background] Bove A, Bongarzoni G, Palone G, Di Renzo R, Di Nicola M, Corradetti L, Corbellini L. Comparative study of an electrothermal bipolar vessel sealing system (LigaSure(R)), a harmonic curved shears (Harmonic Focus), and traditional technique in total thyroidectomy. Am Surg. 2010 Jul;76(7):E94-6. No abstract available. PMID 21683011
- [Background] Siperstein AE, Berber E, Morkoyun E. The use of the harmonic scalpel vs conventional knot tying for vessel ligation in thyroid surgery. Arch Surg. 2002 Feb;137(2):137-42. doi: 10.1001/archsurg.137.2.137. PMID 11822946
- [Background] Yildirim O, Umit T, Ebru M, Bulent U, Belma K, Betul B, Mete D, Omer C. Ultrasonic harmonic scalpel in total thyroidectomies. Adv Ther. 2008 Mar;25(3):260-5. doi: 10.1007/s12325-008-0024-z. PMID 18324377
- [Background] Prgomet D, Janjanin S, Bilic M, Prstacic R, Kovac L, Rudes M, Katic V. A prospective observational study of 363 cases operated with three different harmonic scalpels. Eur Arch Otorhinolaryngol. 2009 Dec;266(12):1965-70. doi: 10.1007/s00405-009-0954-3. Epub 2009 Mar 24. PMID 19308436
- [Background] Sartori PV, De Fina S, Colombo G, Pugliese F, Romano F, Cesana G, Uggeri F. Ligasure versus Ultracision in thyroid surgery: a prospective randomized study. Langenbecks Arch Surg. 2008 Sep;393(5):655-8. doi: 10.1007/s00423-008-0386-3. Epub 2008 Jul 22. PMID 18648850
- [Background] Voutilainen PE, Haglund CH. Ultrasonically activated shears in thyroidectomies: a randomized trial. Ann Surg. 2000 Mar;231(3):322-8. doi: 10.1097/00000658-200003000-00004. PMID 10714624
- [Background] Morton RP, Whitfield P, Al-Ali S. Anatomical and surgical considerations of the external branch of the superior laryngeal nerve: a systematic review. Clin Otolaryngol. 2006 Oct;31(5):368-74. doi: 10.1111/j.1749-4486.2006.01266.x. PMID 17014444
- [Background] Ozlugedik S, Acar HI, Apaydin N, Tekdemir I, Elhan A, Comert A. Surgical anatomy of the external branch of the superior laryngeal nerve. Clin Anat. 2007 May;20(4):387-91. doi: 10.1002/ca.20399. PMID 17022029